CLINICAL TRIAL: NCT01442168
Title: A Phase I/II, Randomized, Open Label, Active Control, Parallel Assignment, Safety/Efficacy Study of Sevuparin/DF02, as an Adjunctive Therapy in Subjects Affected With Uncomplicated Falciparum Malaria
Brief Title: Sevuparin/DF02 as an Adjunctive Therapy in Subjects Affected With Uncomplicated Falciparum Malaria
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Modus Therapeutics AB (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sevuparin/DF02_TSM02
Record Dates: First submitted 2011-09-23; First posted 2011-09-28 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Malaria, Falciparum
Keywords: Uncomplicated Falciparum Malaria; Plasmodium falciparum; Antimalarial treatment; Sevuparin/DF02; Adjuvant therapy; Malanil; Peripheral blood parasitemia; Rosette formation; Maximum tolerated dose
MeSH Terms: conditions — Malaria, Falciparum | interventions — Atovaquone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevuparin/DF02 (Experimental): Sevuparin/DF02 plus anti-malarial regimen (Malanil®)
  Interventions: Drug: Sevuparin sodium + atovaquone/proquanil
- Control (Active Comparator): Anti-malarial regimen (Malanil®) alone
  Interventions: Drug: atovaquone/proquanil

INTERVENTIONS:
Drug: Sevuparin sodium + atovaquone/proquanil — Sevuparin 4 times per day and malanil according to label
  Arms: Sevuparin/DF02
Drug: atovaquone/proquanil — malanil according to label
  Arms: Control

SUMMARY:
The purpose of this study is to determine the tolerability and pharmacokinetics of Sevuparin/DF02 when administered as an i.v. infusion in combination with Malanil® (atovaquone/proguanil) as anti-malarial treatment in subjects affected with uncomplicated malaria. The study will also assess the potential of Sevupatin/DF02 to reduce infected erythrocyte sequestration and rosette formation.

The study consists of a dose escalation part (part 1) followed by an open labelled, randomized comparison of treatment with Sevuparin/DF02 and Malanil® versus Malanil® alone (part 2).

ELIGIBILITY:
Inclusion Criteria:

* Presence of acute uncomplicated P. falciparum malaria, confirmed by positive blood smear with asexual forms of a single species (P. falciparum)
* Counts of asexual forms of P. falciparum: 10 000- 100 000/ul with or without gametocytaemia
* Presence of fever defined as > 38°C tympanic temperature or a history of fever within the last 24 hours

Exclusion Criteria:

* Mixed infection with other Plasmodium species
* Any criteria of severe or complicated malaria as defined by the WHO, 2010
* Use of high doses aspirin (more than 100 mg/day) or dual anti-platelet therapy or use of heparin,Low Molecular Weight Heparin (LMWH) or warfarin
* Presence of significant anemia as defined by Hb <8 g/dL or Hct < 25%
* A platelet count < 50,000/μL
* Presence of febrile conditions caused by diseases other than malaria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities according to specified criteria | During treatment and 14 days post treatment follow-up.
Area under the curve of late stage peripheral blood parasitemia over time (Part 2). | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anna Leitgeb, PhD, Study Director — Modus Therapeutics AB
Locations (3):
- Thailand (3):
  - Mae Ramat Hospital, Mae Ramat, Changwat Tak
  - Maesot General hospital, Mae Sot, Changwat Tak
  - Hospital for Tropical Diseases, Bangkok

REFERENCES:
- [Derived] Leitgeb AM, Charunwatthana P, Rueangveerayut R, Uthaisin C, Silamut K, Chotivanich K, Sila P, Moll K, Lee SJ, Lindgren M, Holmer E, Farnert A, Kiwuwa MS, Kristensen J, Herder C, Tarning J, Wahlgren M, Dondorp AM. Inhibition of merozoite invasion and transient de-sequestration by sevuparin in humans with Plasmodium falciparum malaria. PLoS One. 2017 Dec 15;12(12):e0188754. doi: 10.1371/journal.pone.0188754. eCollection 2017. PMID 29244851